CLINICAL TRIAL: NCT00723359
Title: A Phase I Dose Escalation Study to Evaluate Maximum Tolerated Dose (MTD), Pharmacokinetics (PK), and Safety of BT062 in Subjects With Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Safety and Dose Determining Study of BT062 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotest Pharmaceuticals Corporation (Industry)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 969
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Refractory; Relapsed
MeSH Terms: conditions — Multiple Myeloma; Recurrence

ARMS (1):
- BT062 (Experimental): BT062 single agent dose escalation
  Interventions: Drug: BT062

INTERVENTIONS:
Drug: BT062 — biologic

SUMMARY:
This Phase I research study is to test the effects (good and bad) and best dose of BT062 in treating patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active multiple myeloma according to the International Myeloma Working Group diagnostic criteria
* Relapsed or relapsed/refractory multiple myeloma
* Previous treatment with both an immunomodulator and a proteosome inhibitor therapy
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (Zubrod) ≤ 2
* Ability to understand and willingness to sign a written informed consent document
* Ability to adhere with the study visit schedule and other protocol procedures
* Life expectancy of ≥ 12 weeks
* Normal organ and marrow function

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C)prior to day 1 or those who have not recovered from AEs due to agents administered more than 3 weeks earlier
* Treatment with another investigational agent during the study or within 4 weeks before day 1
* Major surgery within 4 weeks before day 1 (this does not include placement of vascular access device or tumor biopsies)
* Antineoplastic therapy with biological agents within 2 weeks before day 1
* HAHAs, HACAs, or HAMAs in response to previous MAb therapy
* Previous participation in this study
* Malignancy within 3 years before day 1, excluding treated non-melanoma skin cancer, superficial bladder cancer and carcinoma in-situ of the cervix
* Severe diseases of skin, colon, esophagus, or eye within 1 year before day 1, as judged by the Investigator
* Severe infections necessitating use of antibiotics
* Clinically relevant active infection including active hepatitis B or C or human immunodeficiency virus (HBV, HCV, or HIV) or any other concurrent disease which,in the judgment of the investigator, would make the subject inappropriate for enrollment into this study
* Acute or relevant abnormalities in electrocardiogram (ECG), as judged by the Investigator
* Significant cardiac disease such as recent myocardial infarction (≤ 6 months prior to day 1), unstable angina, uncontrolled congestive heart failure, uncontrolled hypertension, (recurrent or persistent increases in systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≥ 110 mm Hg), uncontrolled cardiac arrhythmias, grade 3 or greater cardiac toxicity from prior chemotherapy
* History of clinically significant drug or alcohol abuse
* Unwillingness or inability to adhere to the requirements of the study
* Concomitant therapy with corticosteroids (except as indicated in low dose for other medical conditions such as inhaled steroid for asthma, or as premedication for administration of certain medications or blood products and for treatment of infusion reactions if needed)
* Concomitant antineoplastic therapies including chemotherapy, radiotherapy, or biological agents during the study
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he or she are included in the study
* Pregnant or breast-feeding
* Unwillingness to use an effective contraceptive method during the study and at least 3 months after administration of study drug - unless subject is naturally infertile. (Acceptable contraceptive methods include oral or injectable contraceptives, intrauterine devices (IUD), double-barrier method, contraceptive patch, surgical sterilization, or condoms.)
* Positive serum or urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | On a weekly basis for the duration of the study
Maximum tolerated dose | About every 2 months for the duration of the study

SECONDARY OUTCOMES:
Qualitative and quantitative toxicities | On a weekly basis for the duration of the study
Pharmacokinetics | On a weekly basis for the duration of the study
Anti-tumor activity | At the beginning of each treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C. Anderson, MD, Study Director — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York